CLINICAL TRIAL: NCT06626126
Title: Efficacy of Lipid-Lowering Therapy Based on Apolipoprotein B Versus LDL-Cholesterol Levels in Patients Undergoing Percutaneous Coronary Intervention: a Multicenter, Randomized Controlled Trial
Brief Title: Efficacy of Lipid-Lowering Therapy Based on Apolipoprotein B Versus LDL-Cholesterol Levels in Patients Undergoing Percutaneous Coronary Intervention
Acronym: ApoB-guidedLLT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Collaborators: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Vu Hoang Vu, Head of Interventional Cardiology Department, PhD MD, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ApoBguidedLLT
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Coronary Arterial Disease (CAD); Percutaneous Coronary Intervention; LDL-cholesterol; Lipid Metabolism Disorders
Keywords: ApoB-guidedLLT; PCI; Coronary artery disease; lipid lowering therapy
MeSH Terms: conditions — Lipid Metabolism Disorders; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LDL-C guided-LLT (Active Comparator): Patients in this group will receive treatment regimens adjusted accordingly to meet the LDL-C targets.
  Interventions: Other: LDL-C-guided-LLT
- ApoB-guided-LLT (Experimental): Patients in this group will receive treatment regimens adjusted accordingly to meet the Apolipoprotein B targets.
  Interventions: Other: ApoB-guided-LLT

INTERVENTIONS:
Other: ApoB-guided-LLT — Patients in this group will receive treatment regimens adjusted accordingly to meet the Apolipoprotein B targets
  Arms: ApoB-guided-LLT
Other: LDL-C-guided-LLT — Patients in this group will receive treatment regimens adjusted accordingly to meet the LDL-C targets.
  Arms: LDL-C guided-LLT

SUMMARY:
This multicenter randomized trial is designed to assess the efficacy of lipid-lowering therapy in patients undergoing percutaneous coronary intervention, comparing an Apolipoprotein B-targeted approach with a Low-Density Lipoprotein Cholesterol (LDL-C)-targeted approach. The primary outcomes are to evaluate the proportion of patients achieving lipid-lowering treatment goals at the 1-year follow-up between the two treatment strategies: Apolipoprotein B-based therapy versus LDL-C-based therapy.

DETAILED DESCRIPTION:
This multicenter randomized trial is designed to assess the efficacy of lipid-lowering therapy in patients undergoing percutaneous coronary intervention, comparing an Apolipoprotein B-targeted approach with a Low-Density Lipoprotein Cholesterol (LDL-C)-targeted approach. The primary outcomes are to evaluate the proportion of patients achieving lipid-lowering treatment goals at the 1-year follow-up between the two treatment strategies: Apolipoprotein B-based therapy versus LDL-C-based therapy.

All patients with coronary artery diseases with PCI agreeing to participate will be included. Patient data will be collected and managed through REDCap. These data include information of patient demographics, clinical history and presentations, treatments, and blood test results. The data collection forms are based on EUROHEART data set.

After undergoing percutaneous coronary intervention with drug-eluting stents, participants will be randomly allocated to one of two groups:

1. Patients managed with lipid-lowering therapy targeting LDL-C levels
2. Patients managed with lipid-lowering therapy targeting Apolipoprotein B levels Follow-up assessments will take place at 1, 2, 6, and 12 months post-discharge. During these outpatient visits, a full lipid profile will be performed, including total cholesterol, LDL-C, HDL-C, triglycerides, and Apolipoprotein B. Treatment regimens will be adjusted accordingly to meet the respective targets: LDL-C below 55 mg/dL or Apolipoprotein B below 65 mg/dL.

Moreover, the study aims to assess the incidence of major cardiovascular events, such as all-cause mortality, myocardial infarction, target vessel revascularization, and stroke, at the 1-year follow-up. These outcomes will be compared between the two groups to evaluate the efficacy of Apolipoprotein B-targeted therapy versus LDL-C-targeted therapy in achieving lipid-lowering goals.

The data will be entered into the REDCap program, which will subsequently be processed with the R 4.1.0 program. With a p value < 0.05 and a 95 percent confidence interval, all of the analyses are statistically significant. The investigators employ descriptive statistics, one-variable statistics, and statistics with multiple variables. Qualitative data will be presented as rates and percentages using descriptive statistics, the data will then be processed using the Chi-square test. The investigators report quantitative data as mean (standard deviation) for normal distributions and median (interquartile range) for other distributions. The investigators will use an unpaired t-test to compare means.

Primary Outcome Measures To evaluate the therapeutic efficacy of lipid-lowering therapy predicated on target Apolipoprotein B or target Low-Density Lipoprotein Cholesterol (LDL-C) levels at the one-year follow-up in patients undergoing percutaneous coronary intervention (PCI). Specifically, the primary objective is to conduct a comparative analysis of the achievement rates of lipid-lowering therapeutic targets at the one-year in PCI patients between two cohorts: one receiving therapy tailored to Apolipoprotein B targets versus another receiving treatment based on LDL-C targets.

Secondary Outcome Measures

1. To evaluate the comparative effectiveness of lipid-lowering therapies guided by Apolipoprotein B or LDL-C target levels at the one-year follow-up in post-PCI patients, with a particular focus on comparing the incidence of major adverse cardiovascular events (MACE), including all-cause mortality, myocardial infarction, target vessel revascularization, and stroke, between the two treatment groups: one group managed to Apolipoprotein B targets and the other to LDL-C targets.
2. To compare the incidence and severity of adverse drug reactions (ADRs) associated with lipid-lowering therapies between the two study groups at the one-year follow-up, with one group managed to Apolipoprotein B targets and the other managed to LDL-C targets.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older.
2. Patients undergoing percutaneous coronary intervention (PCI) with drug-eluting stents (DES).
3. Patients who agree to participate and provide informed consent.

Exclusion Criteria:

1. Inability to Provide Informed Consent: Patients who are unable or unwilling to provide consent.
2. Limited life expectancy: patients with a life expectancy of less than 12 months due to other non-cardiac conditions.
3. Liver Disease: patients with cirrhosis or significant liver dysfunction.
4. Patients with contraindication to statin or other lipid-lowering therapy.
5. Any condition that may interfere with the study process, including treatment adherence or follow-up appointments (e.g., dementia, alcohol abuse, severe debilitation, long distances required for follow-up, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1448 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of lipid-lowering therapy predicated on target Apolipoprotein B or target Low-Density Lipoprotein Cholesterol (LDL-C) levels | 1 year
  To evaluate the therapeutic efficacy of lipid-lowering therapy predicated on target Apolipoprotein B or target Low-Density Lipoprotein Cholesterol (LDL-C) levels at the one-year follow-up in patients undergoing percutaneous coronary intervention (PCI). Specifically, the primary objective is to conduct a comparative analysis of the achievement rates of lipid-lowering therapeutic targets at the one-year in PCI patients between two cohorts: one receiving therapy tailored to Apolipoprotein B targets versus another receiving treatment based on LDL-C targets.

SECONDARY OUTCOMES:
Effectiveness of lipid-lowering therapies guided by Apolipoprotein B or LDL-C target levels at the one-year follow-up in post-PCI patients, with a particular focus on comparing the incidence of major adverse cardiovascular events (MACE) | 1 year
  To evaluate the comparative effectiveness of lipid-lowering therapies guided by Apolipoprotein B or LDL-C target levels at the one-year follow-up in post-PCI patients, with a particular focus on comparing the incidence of major adverse cardiovascular events (MACE), including all-cause mortality, myocardial infarction, target vessel revascularization, and stroke, between the two treatment groups: one group managed to Apolipoprotein B targets and the other to LDL-C targets.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No